CLINICAL TRIAL: NCT03857139
Title: The Impact of Opioid Misuse on Tobacco Smoking Cessation
Brief Title: Opioids and Smoking Cessation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Grant funding not obtained
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Andrew Rogers, Principal Investigator, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001467
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Smoking; Smoking Cessation; Smoking, Tobacco; Opioid Use; Opioid Abuse
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Smoking; Opioid-Related Disorders | interventions — Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NRT smoking Cessation Intervention (Experimental): All participants will be provided with the Nicotine Patch as an intervention
  Interventions: Drug: Nicotine patch

INTERVENTIONS:
Drug: Nicotine patch — Participants will receive the transdermal nicotine patch (TNP) to use during the first 2 weeks post-quit. We chose the TNP because of the extensive empirical literature supporting its effectiveness and safety, ease of use, and relatively benign side effect profile. Anxiety and depressive symptoms predict poor smoking cessation outcomes among individuals receiving NRT , suggesting that emotional disturbance influences relapse even in the context of NRT.
  Other Names: Nicotine Replacement Therapy; Transdermal Nicotine Patch

SUMMARY:
The selection hypothesis of smoking prevalence posits that smokers who are not able to quit successfully are "burdened" by specific characteristics that make it more challenging to quit1. For example, those less successful in quitting smoking may be more nicotine dependent or more likely to suffer from substance use, psychiatric, or medical conditions. In line with this perspective, smoking prevalence has stabilized in the US, presumably because the remaining population has become increasingly representative of those "at-risk smokers" who are unable to quit2. Emerging evidence suggests that persons who suffer from opioid misuse, defined as opioid use without a prescription, at a dose or frequency higher than prescribed, or for a non-medical purpose (e.g., getting high),3 may constitute such a high-risk group. Opioid misuse affects greater than 16% adults who use opioids4 and up to 29% of those with chronic pain.5 The prevalence of tobacco smoking in this group may exceed twice that observed in the general population, and smokers misusing opioids are almost twice as likely to be dependent on nicotine6,7. Yet, the role of opioid misuse in periods of early abstinence and smoking cessation has yet to be explored. The main objective of the present proposal is to fill existing gaps in knowledge by examining the extent to which opioid misuse is associated with decreased success during early smoking abstinence and over the course of an attempt to quit smoking, and to identify mediators and moderators of opioid-smoking relations in this context. This contribution is clinically-significant from a public health standpoint because it will directly guide the development of novel psychosocial/behavioral smoking cessation interventions to help this high-risk population of smokers quit by targeting unique vulnerability processes that result in poor cessation outcomes.

DETAILED DESCRIPTION:
B. BACKGROUND/SIGNIFICANCE B.1. Tobacco Smoking. Smoking is responsible for over 40% of premature deaths and disability in the US1, and has been estimated to cost $96 billion in direct medical expenses and $97 billion in lost productivity each year12. Although over 40% of the 48 million Americans that still smoke make a serious quit attempt each year, either on their own (i.e., self-guided quit) or with assistance from formal treatment, less than 5% are able to abstain from smoking for greater than 3 months9. The selection hypothesis of smoking prevalence posits that smokers who are not able to quit successfully are "burdened" by specific characteristics that make it more challenging to quit13. For example, those less successful in quitting smoking may be more nicotine dependent or more likely to suffer from substance use, psychiatric, or medical conditions. According to this perspective, smoking prevalence should begin to stabilize as the remaining population becomes increasingly representative of those "at-risk smokers" who are unable to quit1. There is consensus that significant populations of at-risk adult smokers are present in the general population2. Yet, there remains little understanding of the subgroups of "at-risk smokers" and the processes governing relapse among them14. Emerging evidence suggests that smokers who suffer from opioid misuse may constitute such a "high-risk group"15,16.

B.2. Prevalence of Comorbid Opioid Misuse and Tobacco Smoking. Like smoking, opioid misuse, defined as opioid use without a prescription, at a dose or frequency higher than prescribed, or for a non-medical purpose (e.g., getting high)3, is a critical national health problem that burdens over 11.5 million American adults17, with annual direct medical treatment and lost productivity costs in excess of $504 billion17. Opioid misuse often leads to hypervigilance for somatic perturbation, significant emotional distress, physical deconditioning, and functional disability18-20. According to NIH, the deleterious effects of opioid misuse have been demonstrated in morbidity, immune function, sleep, cognition, eating, mobility, and affective distress11. Clinical and epidemiological population estimates indicate that the prevalence of smoking among persons misusing opioids (upwards of 48%21) may be greater than twice the rate (19%) observed in the general population22-24. Daily smokers are 5 times more likely than non-smokers to meet criteria for past year opioid misuse16.

B.3. Complex Interrelations between Opioid Misuse and Tobacco Smoking. Although interrelations between opioid misuse and smoking have been of clinical interest for decades25, research in this area has only begun to develop. Studies provide evidence of covariation between tobacco smoking and the development and maintenance of opioid misuse16. Chronic nicotine exposure may result in dysregulation of the endogenous opioid system, leading to greater somatic perturbation (e.g., pain) and cross-tolerance to prescription opioids26. There is also evidence that nicotine may sensitize the neural system to enhance the rewarding properties of opioid medications27, which is consistent with incentive-sensitization theories of addiction28,29. Although limited, available work has begun to model the interrelations between opioid misuse and tobacco smoking. One recent study using a representative sample, for example, found that smokers were more likely than non-smokers to report past year opioid misuse, as well as meet criteria for opioid use disorder, and these results were evident over and above depression and alcohol use16. Further, initiating tobacco use prior to the age of 14 and reporting greater tobacco dependence were robustly associated with past-year opioid misuse16.

B.4. Limitations of Opioid Misuse-Tobacco Research. Despite the public health importance of the comorbidity between opioid misuse and smoking, there are substantive gaps in extant research and knowledge. Without such knowledge, it is difficult to develop or adapt smoking cessation treatments to meet the needs of this neglected population. First, despite the established association between opioid misuse and smoking16,24, there are no data addressing the impact of opioid misuse on smoking cessation. There is a clear need to develop research to understanding the extent to which opioid misuse may impair successful smoking cessation. To address this gap, the present proposal seeks to test the extent to which opioid misuse interferes with smoking cessation and theoretically and empirically established factors of negative affect states and nicotine withdrawal/craving that occur over the course of a cessation attempt. This limitation impedes the ability to begin to understand the possible linkages between opioid misuse and key affective and drug-state processes. It is unfortunate theoretically and clinically because numerous studies have documented that smokers, especially those with greater degrees of nicotine dependence or higher smoking rates, report negative affect and problematic physical and affective nicotine withdrawal symptoms during quitting30-32.

Second, it is yet unknown what specific processes account for poor smoking cessation outcomes among smokers with opioid misuse. Identifying these processes is important for at least two reasons: (a) understanding of the pathway(s) through which opioid misuse affects smoking cessation outcomes so that we can develop a process-based theoretical model of opioid misuse-smoking cessation relations; and (b) explicating such explanatory mechanisms is essential to translating basic research knowledge about opioid misuse and smoking to advances in specialized behavioral and pharmacologic smoking cessation interventions for smokers misusing opioid33. The present proposal is therefore innovative in exploring mechanisms that affect opioid-smoking linkages.

Third, there is a need to identify possible moderators of smoking-opioid relations. Although many possible moderators exist, comorbid pain is one leading candidate. Symptoms of (current) moderate to severe pain are more prevalent among both smokers and persons misusing opioids16,34, often doubling rates observed in the general population. Among persons with chronic pain, such comorbidity has been associated with overall greater pain intensity and chronicity, increased functional impairment, and reduced pain-treatment efficacy35,36. Theoretically, chronic pain is therefore apt to increase the severity of nicotine withdrawal and craving and decrease quit success, especially among smokers with opioid misuse. Additionally, sex is another potential candidate as a moderator of smoking-opioid relations37. Specifically, females relative to males often report more difficulty quitting smoking,38,39 due in part to holding more positive expectancies for smoking effects on mood and appetite40-42. In terms of opioid misuse, although less is known, females compared to males receive less treatment for opioid misuse43,44 and report more mood disturbances45-47. Theoretically, these data may suggest that sex differences could exist among tobacco smokers with opioid misuse, such that females may have greater difficulty reducing their tobacco use in the context of opioid misuse.

B.5. Integrative Model. Although presently no integrative model of smoking-opioid co-use has been offered, several mechanisms may be involved. Such mechanisms could include genes central to regulating certain brain chemical systems48-50, neurobiological mechanisms involved in the cross-tolerance and cross-sensitization to both drugs51,52; conditioning mechanisms (e.g., craving for opioids or nicotine elicited by certain environmental cues)53, or individual differences in psychosocial factors (e.g., personality characteristics)54. There is highly limited research addressing these mechanisms. Drawing from past work (see B.3.), I have theorized that smokers with opioid misuse, compared to those without, may be more cognitively, affectively, and behaviorally reactive to aversive internal cues (e.g., nicotine withdrawal, negative emotional states) during periods of smoking deprivation. For example, individuals who misuse opioids may be more apt to engage in catastrophic thinking toward these aversive internal cues (e.g., "I cannot tolerate this distress!")55,56 and experience greater change in the intensity of negative affect, nicotine withdrawal symptoms (e.g., more intense restlessness ), and craving (e.g., "I need to smoke now"). As a result, opioid misuse may drive the affective and drug-state experiences (negative affect and withdrawal symptoms) experienced during a quit attempt. Consequently, individuals with misuse opioids may tend to rely on smoking to cope with such aversive internal distress. From this perspective, aversive internal states (negative affect and nicotine withdrawal symptom)57, may mediate the relation between misuse and lapse/relapse to smoking. Further, individual differences factors, such as severity of pain and sex, could moderate opioid-smoking relations.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-65 years of age. 2. Daily smoker (≥ 10 cigarettes per day for at least one year), biochemically confirmed via Carbon Monoxide [CO] analysis at least 8 ppm.

  3. Motivation to quit smoking (≥ 5 on a 0-10 scale) 4. Interested in making a serious quit attempt in the next month 5. Not have decreased number of cigarettes by more than half in the past 6 months 6. Own a smartphone (for EMA) 7. Report of current (past 30-day) opioid use (opioid misuse group) 8. Verification of opioid use by positive urine toxicology screen & Positive Aberrant Drug Behavior Index (opioid misuse group)
* PDUQ > 11, +POTQ, +urine toxicology screen

Exclusion Criteria:

* 1. Current use of psychotropic medication. 2. Current use of nicotine replacement therapy, Zyban, or Chantix (or intention to use).

  3. Use of other tobacco products, including e-cigarettes. 4. Current treatment for opioid misuse, including methadone, buprenorphine, or naltrexone.

  5. Current diagnosis of Opioid Use Disorder. 6. Pregnancy (by self-report) 7. Limited mental capacity or inability to provide informed consent 8. Current suicidality (by structured clinical interview) 9. Lifetime or current psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Point Prevalence Abstinence | 3 months post-quit date
  CO Biochemical Verification of smoking abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Rogers, M.A., Principal Investigator — University of Houston
Locations (1):
- Anxiety and Health Research Laboratory, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No